CLINICAL TRIAL: NCT02042157
Title: Quality of Life in Adults Impaired Functioning - A Randomized Controlled Trial of Bidet vs Usual Toileting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment malfunction.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mark Cullen, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22588
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Toileting in Adults With Impaired Functional Status; Caregiver Burden for Those Who Care for Adults With Impaired Functional Status; UTI in Adults With Impaired Functional Status
Keywords: Quality of Life; Caregivers; Caregiver burden; Urinary Tract Infections; Bidet; Women's health; Toileting; Hygiene; Activities of Daily Living; Functional impairment; Geriatrics
MeSH Terms: conditions — Caregiver Burden; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bidet use (Experimental): This arm will have a bidet installed in their home bathroom and be instructed how to use it. This arm will use the bidet for usual toileting for a period of two years.
  Interventions: Behavioral: Bidet use
- Usual Toileting (Placebo Comparator): This group will toilet as usual.
  Interventions: Other: Regular toileting
- Caregivers of PT in Arm 1 (bidet use) (Experimental): Participants with functional impairment will be randomized into one of two arms (bidet use or usual toileting). Their caregivers will be enrolled and their randomization is "bundled" with the study participant who they care for. This arm will care for participants who have been randomized to bidet.
  Interventions: Behavioral: Bidet use
- Caregivers of PT in Arm 2 (usual toileting) (Placebo Comparator): Participants with functional impairment will be randomized into one of two arms (bidet use or usual toileting). Their caregivers will be enrolled and their randomization is "bundled" with the study participant who they care for. This arm will care for participants who have been randomized to usual toileting.
  Interventions: Other: Regular toileting

INTERVENTIONS:
Behavioral: Bidet use — Participants used a bidet, a device installed on the toilet that provides fresh water to help clean the bottom and genitalia after having a bowel movement or urinating.
  Arms: Bidet use; Caregivers of PT in Arm 1 (bidet use)
Other: Regular toileting — Patients in the control arm will toilet as usual.
  Arms: Caregivers of PT in Arm 2 (usual toileting); Usual Toileting

SUMMARY:
Our expectations (hypotheses) are:

Primary outcome

1. Regular bidet use will improve quality of life around elimination in adults with impaired functional status. Functional status will be measured by activities of daily living (ADL).
2. Regular bidet use by adults with impaired functional status will improve the quality of life around toileting for their caregivers.

   Secondary
3. Regular bidet use will reduce the incidence, frequency and severity of constipation (as measured by self-report) in adults with impaired functional status.
4. Regular bidet use will reduce the incidence of urinary tract infection (UTI) in adult women with impaired functional status.

DETAILED DESCRIPTION:
The study will assess the use of a bidet (a device that is attached to the toilet which allows a person to wash their genitalia after elimination) in improving toilet related quality of life for functionally impaired individuals as measured by ADLs and caregivers of functionally impaired adults. We also want to see if bidet use is effective in lowering the incidence of urinary tract infections in this high risk population.

Functional impairment around toileting has been shown to negatively impact quality of life (QOL) for both patients and their caregivers. We hope to learn if the use of bidet will improve QOL in this population.

Urinary tract infections increase the risk of morbidity and mortality in women with impaired functional status. Specifically the risk of hospitalization, sepsis, kidney failure and other complications. There are not currently effective forms of non-pharmaceutical prevention. Bidets are safe, inexpensive and hygienic. Individuals with functional impairment often have difficulty maintaining their hygiene due to frailty and functional limitations. It is our hope that addressing these issues will lead to a reduced incidence of UTI.

Constipation is a common problem in elderly adults and in adults with impaired functional status. It is our hope that the bidet will reduce the frequency and severity of constipation (as measured by self report).

ELIGIBILITY:
Inclusion Criteria:

Sample 1 (adults with impaired functional status):

Age: 55-95 Sex: Female Ethic background: Reflecting the population at Stanford Hospital and Clinics who meet the inclusion criteria and who agree to participate.

Sample 2 (caregivers of participants in Sample 1) Adults over the age of 21 caring for an adult with impaired functional status who has enrolled in this randomized controlled trial. Sex and ethnic background will reflect the demographic of the caregivers for the population in Sample 1.

Exclusion Criteria:

Participants not meeting the inclusion criteria.

Additional exclusion criteria:

1. Life expectancy less than 2 years
2. The inability to read and write English.
3. Patients with indwelling urinary (e.g. Foley) catheters
4. Use of any water based cleaning system after toileting at home in the past 12 months (bidet, water pot, douche etc).
5. Fully incontinent (eg diaper use)
6. Moderate to severe cognitive impairment (15 or lower on the MOCA)

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Improved quality of life as measured QoL questionnaire | 24 months
  We are measuring the quality of life using a validated QoL questionnaire which has been slightly modified to include questions around toileting.
Caregiver burden for caregivers of adults with functional limitations as measured by a validated caregiver burden questionnaire. | 24 months
  We will measure caregiver burden using a validated instrument.

SECONDARY OUTCOMES:
Incidence of UTI as measured by enquiry and chart review (female patients only). | 24 months
  Every month we will screen female patients in both arms of the study to ask them if they have had any symptoms of UTI or sought medical attention for UTI.
  We will also review their chart for diagnosis of UTI or prescription of a medication for UTI. Either self-report of a diagnosis or prescription for a medication of a UTI or a report of UTI in the chart will be considered an incidence of UTI.
Incidence of constipation as measured by self report | 24 months
  We will ask patients on a monthly basis if they have had constipation.
Severity (measured by self report) of constipation | 24 months
  For those patients who report having had constipation, will ask them to rate the severity of their constipation on a monthly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Yusra Hussain, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- See also: Search engines for all clinical research taking place at Stanford Medical Center — http://med.stanford.edu/clinicaltrials/
- See also: Portal for Stanford Aging Adult Services — http://stanfordhospital.org/forPatients/patientServices/agingAdults/